CLINICAL TRIAL: NCT06810310
Title: Psilocybin: Capturing Brain Mechanisms of Motivation and Neurocognition in Individuals With Opioid Use Disorder
Brief Title: Psilocybin on Brain Mechanisms of Motivation in OUD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anna Rose Childress, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Anna Rose Childress, Ph.D., Research Associate Professor, Department of Psychiatry, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 857697
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose psilobyin (Active Comparator): 1 mg PEX010 capsule, single dose
  Interventions: Drug: psilocybin (low dose)
- High dose psilocybin (Experimental): 25 mg PEX010 capsule, single dose
  Interventions: Drug: Psilocybin (high dose)

INTERVENTIONS:
Drug: Psilocybin (high dose) — PEX010 is the psilocybin produced by Filament
  Arms: High dose psilocybin
Drug: psilocybin (low dose) — 1mg psilocybin, produced by Filament
  Arms: Low dose psilobyin

SUMMARY:
The goal of this study is to test addiction-related brain circuitry (motivation/reward and inhibition) as well as neurocognitive circuitry prior to and following low or high dose psilocybin (PEX010 from Filament). Using fMRI, we will examine brain circuits relevant to drug relapse as well as neurocognitive flexibility circuits in individuals with opioid use disorder.

We will randomize 24 males and females, aged 18 - 60, in the greater Philadelphia area, to either 1mg or 25 mg of psilocybin. Participants will

1. come to our offices for screening visits - these are assessments, interviews, and some medical tests (such as a history and physical, as well as a fasting blood draw) to help us determine eligibility for our study.
2. If not already in an inpatient setting, participants be admitted to an inpatient program for the duration of the psilocybin phases - about two weeks. During this time, they will be brought to our offices at 3535 Market Street in Philadelphia for about 7 visits. These visits include pre-dose psilocybin preparation therapy, baseline assessments and neuropsychological testing, psilocybin dosing, post dose therapy visits, and post dose assessments.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document voluntarily signed and dated by the subject.
* Voluntary enrollment in the residential addiction treatment facility
* Intention on residing within residential addiction treatment facility for the duration of the Pre/Post PSI dosing period.
* Either 1) have a confirmed prescription for BUP-NX in a drug monitoring program database, have been on a stable dose of BUP-NX for at least one week, and plan to continue taking BUP-NX for at least 12 weeks or 2) have received an injection of Sublocade® within the past month, or 3) are currently on methadone maintenance therapy and on a consistent dose for at least a week. Subject must provide a urine that is buprenorphine-positive (for subjects taking buprenorphine) or methadone-positive (for subjects taking methadone), during screening.
* Physically healthy males and females, aged 18-60 years old, who meet criteria for opioid use disorder (based on DSM-5 criteria) as their primary diagnosis and are voluntarily seeking treatment.
* Females must be non-pregnant and non-lactating. Additionally, for females with childbearing potential (i.e., have not undergone sterilization via hysterectomy, bilateral tubal ligation, or bilateral oophorectomy, or at least 1 year post-menopausal) participants must agree to use an acceptable form of contraception (e.g. abstinence, intrauterine device, hormonal injection, hormonal implant, hormonal patch/ring/pill, condoms (male or female), etc.) during study participation and to continue its use for the duration of the study
* Subject must read at or above eighth grade level and speak, understand, and write in English.
* IQ score of greater than or equal to 80.

Exclusion Criteria:

* Participation in clinical trial and receipt of investigational drug(s) during 30 days prior to the research study, except as explicitly approved by the Principal Investigator.
* Currently meets DSM-5 criteria for moderate to severe substance use disorder for any substance other than cocaine, alcohol, marijuana or nicotine as determined by the semi-structured interview. Any prior use of psilocybin is exclusionary. Patients with comorbid Alcohol Use Disorder will be accepted if their alcohol use disorder is not severe enough to require a medicated alcohol detoxiﬁcation.
* Meets current or lifetime DSM-5 criteria for schizophrenia or any psychotic disorder, or organic mental disorder or has a first-degree family history of these disorders, this includes a history of hallucinogen-persistent perception disorder (HPPD)
* Meets current DSM-5 criteria for bipolar disorder

  --Meets current DSM-5 criteria for severe Major Depressive Disorder (mild and moderate MDD as well as in stable remission are allowed if no suicidal risk and no ongoing antidepressant therapy).
* Current or past significant trauma exposure with elevated Post-Traumatic Stress symptoms at the discretion of the PI.
* Presence of any another psychiatric disorder that in the opinion of the PI will interfere with completion of the study or place the patient at heightened risk through participation in the study.
* Current or past month active suicidal ideations or lifetime history of serious suicidal attempt.
* Has evidence of signiﬁcant hepatocellular injury as evidenced by elevated bilirubin levels (greater than 1.3), or, pulmonary (e.g., COPD), endocrine, cardiovascular, renal (creatinine clearance less than or equal to 60ml/min) or gastrointestinal disease (e.g., Crohn's disease), or current HIV infection, and/or clinically signiﬁcant levels (over 3.5x upper limit of normal) of aspartate aminotransferase (AST), and serumalanine aminotransferase (ALT). Patients with documented Gilbert's syndrome will be included regardless of bilirubin levels.
* History of serious head trauma or injury causing loss of consciousness that lasted more than 3 minutes and/or associated with skull fracture or intracranial bleeding or abnormal MRI.
* Seizure disorder or history of seizures not related to drug or alcohol withdrawal (excluding childhood febrile seizure).
* Presence of magnetically active prosthetics, plates, pins, broken needles, permanent retainer, bullets, etc. in patient's body (unless a radiologist conﬁrms that its presence is unproblematic). An x-ray may be obtained to determine eligibility.
* Claustrophobia or other medical condition that disables the participant from lying in the MRI for approximately 60 minutes.
* Non-removable skin patches, at discretion of PI.
* Has received medication that could interact adversely with psilocybin within the time of administration of study agent based on the Medical Director's guidance.
* Needs treatment with any psychoactive (e.g., anti-depressants) medications (with the exception of Benadryl used sparingly, if necessary, for sleep).
* *Have the following cardiovascular conditions:

  1. coronary artery disease, congenital long QT syndrome (prior diagnosis), cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction (prior diagnosis);
  2. tachycardia (deﬁned as heart rate greater than 100 beats per minute);
  3. a clinically signiﬁcant Screening ECG abnormality (e.g., atrial ﬁbrillation); Note: A QTcF interval greater than 450 milliseconds is considered a clinically signiﬁcant ECG abnormality
  4. artiﬁcial heart valve;
  5. any other signiﬁcant current or history of cardiovascular condition, based on the clinical judgment of Medical Director, that would make a participant unsuitable for the study.
* *At Screening or Baseline have elevated blood pressure as deﬁned as:

  1. Screening blood pressure SBP greater than135 mmHg or DBP greater than 85 mmHg on three separate readings; or
  2. Baseline blood pressure SBP greater than140 mmHg or DBP greater than 90 mmHg on three separate readings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Brain measure of GO domain | One week pre dose and one week post dose
  Using fMRI, we will measure the brain response to 500ms evocative cues and 6 second drug-related videos that trigger drug desire
Behavioral measure of GO domain | One week pre dose and one week post dose
  Using a the Affect Bias behavioral task, we will measure the affective bias to opioid and other evocative visual cues.

SECONDARY OUTCOMES:
Brain measure of STOP domain | weeks 1 through 8 (outcomes phase)
  Using fMRI, we will measure the brain response during an Affect-congruent Go-NoGo task, and during 6 second videos with instruction to "Reduce your response to the video by considering the negative consequences of acting on your craving."
Behavioral measure of STOP domain | One week pre dose and one week post dose
  Using a standard behavioral Go0NoGo task, we will measure errors of commission.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No